CLINICAL TRIAL: NCT04123652
Title: Ambulatory Infusions of Lidocaine and Ketamine for Management of Chronic Pain: an Observational Prospective Study
Brief Title: Ambulatory Infusions of Lidocaine and Ketamine for Management of Chronic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allevio Pain Management Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16124-11:10:3610-082018
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2017-11

CONDITIONS: Chronic Neuropathic Pain and Fibromyalgia
Keywords: Neuropathic pain; Fibromyalgia; Lidocaine infusion; Ketamine infusion; Chronic pain
MeSH Terms: conditions — Fibromyalgia; Neuralgia; Chronic Pain | interventions — Lidocaine; Ketamine

STUDY DESIGN:
Intervention Model Description: Patients are assessed for eligibility on their first visit (screening visit); additional visits may be required to address patient questions and collect baseline data. Qualified participants will be scheduled for their 5 infusions at 8 week intervals.
  Dosing and infusion orders are completed by one of the physician-investigators prior to patient arrival based on body weight, and modified if required after individual evaluation. Based on published literature and clinical impression, higher doses seem to be more effective and result in longer pain relief. Therefore, subsequent infusion doses will be increased to the maximally tolerated doses (i.e. minimal side effects).
  Participants will be asked to complete the follow-up questionnaires every four weeks starting from their first infusion up to 8 times. On their last study visit, 4 weeks following the last infusion, participants will have an exit interview in addition to completing study measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lidocaine and ketamine infusion (Other)
  Interventions: Drug: Lidocaine Hydrochloride 2% Intravenous Solution, DIN 02421992

INTERVENTIONS:
Drug: Lidocaine Hydrochloride 2% Intravenous Solution, DIN 02421992 — An intravenous will be started. • Lidocaine - initial dose of 5.0 mg/kg +/- 1.0 mg/kg (based on actual weight, up to maximum dose 600 mg) over 45 minutes, followed by increases of 0.5 mg/kg each infusion based on tolerability of side effects, not to exceed 7 mg/kg or 600 mg.
  • Ketamine - initial dose of 0.1 mg/kg (based on actual weight) over 45 minutes (rounded to nearest 5 mg, up to maximum 15 mg), increased by 0.1 mg/kg (rounded to nearest 5 mg) each infusion based on tolerability of side effects During the infusion patient will be monitored by another MD for BP, PR, PO2. Patients will not be allowed to drive for 24 hours.
  Other Names: ketamine Hydrochloride, Serial# 5751304560, DIN 02246796

SUMMARY:
As lidocaine and ketamine provide analgesia by acting on different molecular pathways, administering them together may produce synergistic effects, which can allow for using a lower dose of each medication and thereby reducing the corresponding side effects. To the investigator's knowledge, despite the common practice of multimodal analgesia, lidocaine-ketamine infusions have never been studied prospectively in an out of hospital setting to treat neuropathic pain. The aim of the present study is to evaluate the effectiveness of the current routine practice of lidocaine-ketamine infusions conducted at Allevio Pain Management Clinic, a large outpatient community based chronic pain management facility. Lidocaine-ketamine infusions are prescribed to patients that have pain that is considered to be neuropathic for which standard anti-neuropathic medications have been ineffective or poorly tolerated by patients. A prospective longitudinal study.

DETAILED DESCRIPTION:
Study objectives

1. To evaluate effectiveness of lidocaine-ketamine infusions in reducing neuropathic pain, as assessed using the Revised Pain Quality Assessment Scale (PQAS-R) and Short Form Brief Pain Inventory (BPI-SF).
2. To evaluate the effects of lidocaine-ketamine infusions on the measures of Global Improvement and Satisfaction Score, Pain Self-Efficacy Questionnaire (PSEQ), Pain Catastrophic Scale (PCS), Beck Depression Inventory (BDI), and Patient self-reported perceived duration of effect (PSPDE).
3. To assess, analyze, and report adverse events

The study will be conducted per IMMPACT recommendations (17). Multi variable parameters will be captured: pain unpleasantness, physical function, emotional function, global improvement and satisfaction with treatment, adverse events and disposition. Additional instruments will be used in the triage process and follow-up (S-LANSS, PSEQ).

Number of subjects: all eligible consecutive patients accepted for lidocaine-ketamine infusions over period of 6 months.

Patients with multi focal and/or non-dermatomal pain with neuropathic component will be included.

Dosing and infusion orders are completed by one of the physician-investigators prior to patient arrival based on body weight, and modified if required after individual evaluation. Based on published literature and clinical impression, higher doses seem to be more effective and result in longer pain relief. Therefore, subsequent infusion doses will be increased to the maximally tolerated doses (i.e. minimal side effects).

Doses will be calculated using the following:

* Lidocaine - initial dose of 5.0 mg/kg +/- 1.0 mg/kg (based on actual weight, up to maximum dose 600 mg) over 45 minutes, followed by increases of 0.5 mg/kg each infusion based on tolerability of side effects, not to exceed 7 mg/kg or 600 mg.
* Ketamine - initial dose of 0.1 mg/kg (based on actual weight) over 45 minutes (rounded to nearest 5 mg, up to maximum 15 mg), increased by 0.1 mg/kg (rounded to nearest 5 mg) each infusion based on tolerability of side effects.

Standard clinic procedure will be followed for completing the infusions and managing side effects. The infusion will be initiated at 360 ml/hour for planned completion in 45 minutes, rate adjusted if side effects develop. Total doses of medication are recorded in the medical record.

Data collection and Management All study tools will be completed by patients online using, or in the clinic RedCap system. RedCap is a mature, secure web application for building and managing online surveys and databases (Vanderbilt University). The system is secured by SSL protocol and data is encrypted. Patients will be contacted via Email with a secure link to RedCap database, or if they would not be able to do it at home research, they can complete the questionnaires with research coordinator's assistant in secure computers at the clinic. Participant will receive reminders about upcoming visits and promoted to complete the follow-up forms. Allevio data protection is also SSL enabled and secured by SHA256, and they are issued by Rapid SSL and purchased through Ceerts4Less.

ELIGIBILITY:
Inclusion Criteria:

Pain duration > 3 months;

Multifocal and/or non-dermatomal neuropathic pain per Pain Diagram;

Failed medical management with at least 2 neuromodulation agents (e.g., gabapentinoids, antidepressants, cannabinoids);

Neuropathic component (12 or more points on S-LANSS);

Exclusion Criteria:

Non-English speakers;

Refusal to sign informed consent;

Allergy to ketamine and/or lidocaine;

Known relative contraindications to ketamine use which include poorly controlled systemic illnesses: hypertension, hyperthyroidism, ischemic heart disease, heart failure, psychiatric comorbidity (e.g., psychosis, schizophrenia, dissociative state);

Known contraindication to lidocaine use which include current symptomatic or clinically significant brady- or tachyarrhythmia, systolic blood pressure <90 or >180 mmHg;

Scheduled interventions targeting neuropathic pain: epidural injections, peripheral nerve blocks, Bier block, radiofrequency of dorsal root ganglia and peripheral nerves, additional lidocaine or ketamine infusions;

Newly added analgesic or neuromodulating medications within 30 days;

Recently performed neuromodulating interventions within 90 days;

Previous lidocaine-ketamine, lidocaine or ketamine infusion within 6 months;

Acute intoxication or active illegal substance abuse;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of effectiveness of lidocaine-ketamine infusions: PQAS-R | 4 weeks after the first infusion and every 4 weeks up to 36 weeks
  Primary outcome measure: relative change on the PQAS-R. Moderate clinically important improvement is considered as 30% reduction (Dworkin et al., 2008)

SECONDARY OUTCOMES:
Effect of lidocaine and ketamine infusion on BDI | Baseline to end-of-study every 4 weeks up to 36 weeks
  Effect of lidocaine and ketamine infusion on Beck's Depression Inventory
Effect of lidocaine and ketamine infusion on PGIC | Baseline to end-of-study every 4 weeks up to 36 weeks
  Effect of lidocaine and ketamine infusion on Pain Global Improvement and Satisfaction
Effect of lidocaine and ketamine infusion on BPI | Baseline to end-of-study every 4 weeks up to 36 weeks
  Effect of lidocaine and ketamine infusion on Brief Pain Inventory
Effect of lidocaine and ketamine infusion on PQAS-R | Baseline to end-of-study every 4 weeks up to 36 weeks
  Effect of lidocaine and ketamine infusion on Revised Pain Quality Assessment Scale
Effect of lidocaine and ketamine infusion on PSEQ | Baseline to end-of-study every 4 weeks up to 36 weeks
  Effect of lidocaine and ketamine infusion on Patient Self-Efficacy Questionnaire
Effect of lidocaine and ketamine infusion on PCS | Baseline to end-of-study every 4 weeks up to 36 weeks
  Effect of lidocaine and ketamine infusion on Pain Catastrophizing Scale
Effect of lidocaine and ketamine infusion on PSPDE | Baseline to end-of-study every 4 weeks up to 36 weeks
  Effect of lidocaine and ketamine infusion on viii. Patient self-reported perceived duration of effect
Effect of lidocaine and ketamine on narcotic consumption | Baseline to end-of-study up to 36 weeks
  Effect of lidocaine and ketamine infusion on narcotic consumption

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Safakish, MD.FRCPC, Principal Investigator — Allevio Pain Management Clinic
Locations (1):
- Allevio Pain Management Clinic, Toronto, Ontario, Canada

REFERENCES:
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Result] BONICA JJ. The management of pain of cancer. J Mich State Med Soc. 1953 Mar;52(3):284-90. No abstract available. PMID 13035388
- [Result] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Result] IASP. (2003). How Prevalent Is Chronic Pain? International Association for the Study of Pain. Retrieved from https://www.iasp-pain.org/files/Content/ContentFolders/Publications2/PainClinicalUpdates/Archives/PCU03-2_1390265045864_38.pdf
- [Result] Goldberg DS, McGee SJ. Pain as a global public health priority. BMC Public Health. 2011 Oct 6;11:770. doi: 10.1186/1471-2458-11-770. PMID 21978149
- [Result] Cho SK, Heiby EM, McCracken LM, Moon DE, Lee JH. Daily functioning in chronic pain: study of structural relations with posttraumatic stress disorder symptoms, pain intensity, and pain avoidance. Korean J Pain. 2011 Mar;24(1):13-21. doi: 10.3344/kjp.2011.24.1.13. Epub 2011 Feb 25. PMID 21390174
- [Result] Wahl AK, Rustoen T, Rokne B, Lerdal A, Knudsen O, Miaskowski C, Moum T. The complexity of the relationship between chronic pain and quality of life: a study of the general Norwegian population. Qual Life Res. 2009 Oct;18(8):971-80. doi: 10.1007/s11136-009-9515-x. Epub 2009 Aug 18. PMID 19688608
- [Result] Gaskin DJ, Richard P. The economic costs of pain in the United States. J Pain. 2012 Aug;13(8):715-24. doi: 10.1016/j.jpain.2012.03.009. Epub 2012 May 16. PMID 22607834
- [Result] Fitzcharles MA, Baerwald C, Ablin J, Hauser W. Efficacy, tolerability and safety of cannabinoids in chronic pain associated with rheumatic diseases (fibromyalgia syndrome, back pain, osteoarthritis, rheumatoid arthritis): A systematic review of randomized controlled trials. Schmerz. 2016 Feb;30(1):47-61. doi: 10.1007/s00482-015-0084-3. PMID 26767993
- [Result] Ballantyne JC, Mao J. Opioid therapy for chronic pain. N Engl J Med. 2003 Nov 13;349(20):1943-53. doi: 10.1056/NEJMra025411. No abstract available. PMID 14614170
- [Result] Noble M, Treadwell JR, Tregear SJ, Coates VH, Wiffen PJ, Akafomo C, Schoelles KM. Long-term opioid management for chronic noncancer pain. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD006605. doi: 10.1002/14651858.CD006605.pub2. PMID 20091598
- [Result] IASP. (1994). Part III: Pain Terms, A Current List with Definitions and Notes on Usage. In Classification of Chronic Pain (second ed., pp. 209-214): IASP Press. Retrieved from
- [Result] van Hecke O, Austin SK, Khan RA, Smith BH, Torrance N. Neuropathic pain in the general population: a systematic review of epidemiological studies. Pain. 2014 Apr;155(4):654-662. doi: 10.1016/j.pain.2013.11.013. Epub 2013 Nov 26. PMID 24291734
- [Result] Campbell, J. N., & Meyer, R. A. (2006). Mechanisms of neuropathic pain. Neuron, 52(1), 77-92. doi:10.1016/j.neuron.2006.09.021 CDC. (2017a). Opioid Overdose. Centers for Disease Control and Prevention. Retrieved from https://www.cdc.gov/drugoverdose/index.html CDC. (2017b). Prescribing Data. Centers for Disease Control and Prevention. Retrieved from https://www.cdc.gov/drugoverdose/data/prescribing.html
- [Result] Gilron I, Watson CP, Cahill CM, Moulin DE. Neuropathic pain: a practical guide for the clinician. CMAJ. 2006 Aug 1;175(3):265-75. doi: 10.1503/cmaj.060146. PMID 16880448
- [Result] Niesters M, Martini C, Dahan A. Ketamine for chronic pain: risks and benefits. Br J Clin Pharmacol. 2014 Feb;77(2):357-67. doi: 10.1111/bcp.12094. PMID 23432384
- [Result] Dale R, Stacey B. Multimodal Treatment of Chronic Pain. Med Clin North Am. 2016 Jan;100(1):55-64. doi: 10.1016/j.mcna.2015.08.012. Epub 2015 Oct 17. PMID 26614719
- [Result] Rogers M, Tang L, Madge DJ, Stevens EB. The role of sodium channels in neuropathic pain. Semin Cell Dev Biol. 2006 Oct;17(5):571-81. doi: 10.1016/j.semcdb.2006.10.009. Epub 2006 Oct 28. PMID 17123847
- [Result] Zhou HY, Chen SR, Pan HL. Targeting N-methyl-D-aspartate receptors for treatment of neuropathic pain. Expert Rev Clin Pharmacol. 2011 May;4(3):379-88. doi: 10.1586/ecp.11.17. PMID 21686074